CLINICAL TRIAL: NCT01967992
Title: Examining the Effects of Diet on Health With an Online Program
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-11813
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; obesity; mindful eating; positive affect; low carbohydrate; ketogenic; diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Obesity | interventions — Diet, Ketogenic; Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- American Diabetes Association recommended diet (Active Comparator): Participants in the American Diabetes Association (ADA) diet group will receive standard ADA advice. The diet includes high-fiber foods (such as vegetables, fruits, whole grains, and legumes), low-fat dairy products, fresh fish, and foods low in saturated fat. They will be asked to use the "plate method" to guide their nutritional choices.
  Interventions: Behavioral: American Diabetes Association Diet
- Low Carbohydrate Diet (Experimental): Participants will be instructed to follow a low carbohydrate, ketogenic diet: carbohydrate intake 20-35 grams a day not including fiber. Foods permitted include: meats, poultry, fish, eggs, cheese, cream, some nuts and seeds, green leafy vegetables, and most other non-starchy vegetables. Because most individuals self-limit caloric intake, no calorie restriction will be recommended.
  Participants will also be taught information about mindfulness and positive affect practices. The mindfulness-based curriculum will focus on the following elements: training on topics such as mindful meditation, mindful eating, awareness of fullness and hunger signals, and taste satiety. The positive emotion curriculum will include: training on topics such as noticing and savoring positive events, gratitude, positive reappraisal, personal strengths, attainable goals, and acts of kindness.
  Interventions: Behavioral: Behavioral: Low Carbohydrate, Ketogenic Diet; Behavioral: Mindfulness and Positive Affect Skills

INTERVENTIONS:
Behavioral: Behavioral: Low Carbohydrate, Ketogenic Diet
  Arms: Low Carbohydrate Diet
Behavioral: American Diabetes Association Diet
  Arms: American Diabetes Association recommended diet
Behavioral: Mindfulness and Positive Affect Skills
  Arms: Low Carbohydrate Diet

SUMMARY:
The study is a pilot, designed to provide data regarding the feasibility and acceptability of conducting such a study on a larger scale. The present study is a randomized controlled clinical trial comparing two programs to help people manage diabetes and lose weight, one using a moderate-carbohydrate diet promoted by the American Diabetes Association (ADA) and the other using on a low-carbohydrate diet (LC) and mindfulness and positive affect lifestyle modifications. Intervention content will include information about nutrition (American Diabetes Association recommended diet or carbohydrate restriction) and, in the LC group, emotion regulation, positive affect, and mindful eating strategies.

DETAILED DESCRIPTION:
Approximately individuals with type 2 diabetes will be randomized in a 1:1 ratio to treatment groups. Classes will occur online. Participants will be evaluated at 0, 16, and 32 weeks. Our main outcome of interest is HbA1c (glycated hemoglobin, a measure indicative of blood glucose levels and tied to diabetes severity).

ELIGIBILITY:
Inclusion Criteria:

1. HbA1c 6.5%-9% at screening.
2. Aged 18 years old and older
3. BMI 25 and above.
4. Willing and able to participate in the interventions such as having sufficient control over their food intake. Must have the ability to make choices about the food they eat; cannot have a lifestyle in which they eat out most of their meals.)

Exclusion Criteria:

1. Unable to provide informed consent.
2. Non English speaker.
3. No current use of insulin, no immediate plans to start or increase diabetic mediations, and no use of diabetes medications besides metformin.
4. A substance abuse, mental health, or medical condition that, in the opinion of investigators, will make it difficult for the potential participant to participate in the intervention. Such conditions may include: cancer, liver failure, unstable coronary artery disease, severe emphysema, binge eating disorder or history of binge eating disorder, bulimia or strong history of bulimia.
5. Previous use or recent changes in medications that can interfere with the measures used in the study: current use of insulin; use of systemic (oral or IV) corticosteroids in the 6 months prior to enrollment or severe autoimmune disorders or other conditions (e.g. rheumatoid arthritis, lupus), that are likely to require these medications; and initiation of new class of psychiatric medications in past 2 months.
6. Pregnant or planning to get pregnant in the next 12 months, breastfeeding or less than 6 months post-partum.
7. Current use of weight loss medications or supplements such as Alli or amphetamine-based drugs that are believed to have some effect on weight.
8. History of or planned weight loss surgery.
9. Vegan or vegetarian. The intervention diets are more challenging for vegan and vegetarian participants.
10. No or very limited internet access at a computer. Must be able to complete the online assessments and access the online class materials.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | baseline to 16 weeks
  We will test whether Hemoglobin A1c changes from pre-intervention to 16 weeks. The key outcome measure will compare the two groups, but we will also assess whether statistically significant changes occur within groups from pre-intervention to 16 weeks.

SECONDARY OUTCOMES:
Hemoglobin A1c | baseline to 32 weeks
  We will test whether Hemoglobin A1c changes from pre-intervention to 32 weeks. The key outcome measure will compare the two groups, but we will also assess whether statistically significant changes occur within groups from pre-intervention to 32 weeks.

OTHER OUTCOMES:
Body weight | baseline to 16 weeks
  We will test whether body weight changes from pre-intervention to 16 weeks. The key outcome measure will compare the two groups, but we will also assess whether statistically significant changes occur within groups from pre-intervention to 16 weeks.
Body weight | baseline to 32 weeks
  We will test whether body weight changes from pre-intervention to 32 weeks. The key outcome measure will compare the two groups, but we will also assess whether statistically significant changes occur within groups from pre-intervention to 32 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Laura R Saslow, PhD, Principal Investigator — University of Michigan; Rick Hecht, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Saslow LR, Mason AE, Kim S, Goldman V, Ploutz-Snyder R, Bayandorian H, Daubenmier J, Hecht FM, Moskowitz JT. An Online Intervention Comparing a Very Low-Carbohydrate Ketogenic Diet and Lifestyle Recommendations Versus a Plate Method Diet in Overweight Individuals With Type 2 Diabetes: A Randomized Controlled Trial. J Med Internet Res. 2017 Feb 13;19(2):e36. doi: 10.2196/jmir.5806. PMID 28193599
- See also: recruitment website for study — http://www.osher.ucsf.edu/research/enroll-in-research-studie/succeed-study/